CLINICAL TRIAL: NCT06258356
Title: Exploring the Use of Remimazolam (BYFAVO®) in Patients at High Risk for ERCP to Reduce Intraoperative Hypotension and Assess Safety and Efficacy: A Randomized Controlled Trial
Brief Title: Remimazolam in High Risk ERCP Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Research Ethic Committee D, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 202310115MIND
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: the Severity and Duration of Intraoperative Hypotension
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Intervention Model Description: One patients receiving Remimazolam, the other patients receiving placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients receiving Remimazolam (Experimental)
  Interventions: Drug: Remimazolam
- patients without Remimazolam (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Remimazolam — novel ultra-short-acting benzodiazepine-like anesthetic.
  Arms: patients receiving Remimazolam
Drug: placebo — normal saline (compared to Remimazolam)
  Arms: patients without Remimazolam

SUMMARY:
We conducted a randomized trial to investigate whether the administration of Remimazolam in patients undergoing high-risk endoscopic retrograde cholangiopancreatography (ERCP) could significantly reduce the occurrence of intraoperative hypotension, facilitate rapid induction, and result in fewer associated complications.

DETAILED DESCRIPTION:
Remimazolam is a novel ultra-short-acting benzodiazepine-like anesthetic used for gastrointestinal endoscopic procedures, characterized by predictable sedation duration and rapid recovery. Propofol, commonly used in clinical practice as an intravenous anesthetic, also exhibits rapid onset, short duration, and quick recovery characteristics. To date, there is relatively limited literature comparing the likelihood of intraoperative hypotension during general anesthesia with these two agents in patients undergoing endoscopic retrograde cholangiopancreatography (ERCP). Additionally, a comparison is needed regarding the frequency of additional sedative doses required during anesthesia induction and the occurrence of major postoperative complications, including pancreatitis.

Therefore, the investigators we conducted a randomized trial to investigate whether the administration of Remimazolam in patients undergoing high-risk ERCP could significantly reduce the occurrence of intraoperative hypotension, facilitate rapid induction, and result in fewer associated complications. The investigators aimed to enroll 60 patients with a 1:1 ratio of ASA III to IV undergoing ERCP. The investigators anticipate that Remimazolam can reduce intraoperative hypotension, acute postoperative pancreatitis, and the occurrence of major organ complications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 20 and 90 years old;
* ASA (American Society of Anesthesiologists) class III to IV;
* Body Mass Index (BMI) between 18 and 30 kg/m².

Exclusion Criteria:

* Uncontrolled hypertension or hypotension, or clinically significant coronary artery atherosclerosis heart disease or heart failure;
* Severe respiratory system disorders;
* Severe sinus bradycardia, heart conduction block, frequent ventricular arrhythmias, or atrial fibrillation;
* Clinically significant coagulation disorders;
* End-stage liver failure or kidney disease requiring dialysis;
* Emergency surgery;
* Peripheral artery disease with upper limb functional impairment;
* Other conditions deemed inappropriate by the investigator, including patients with superficial pharyngeal cancer for whom rapid extubation is not suitable during ERCP.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the duration and severity of hypotension checklist | 1 day (during the ERCP examination)
  during the ERCP examination

IPD SHARING:
Plan to Share IPD: No
due to patients' privacy